CLINICAL TRIAL: NCT00527423
Title: A Randomized, Single-Masked , Long-Term, Safety and Tolerability Study of Intravitreal VEGF Trap-Eye in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: Randomized, Single-Masked, Long-Term, Safety and Tolerability Study of VEGF Trap-Eye in AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VGFT-OD-0702
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Results first posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Macular Degeneration
Keywords: VEGF Trap-Eye; Macular Degeneration; AMD; Neovascular Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) (Experimental)
  Interventions: Drug: VEGF Trap Eye

INTERVENTIONS:
Drug: VEGF Trap Eye — Intravitreal injection
  Other Names: IVT

SUMMARY:
Rollover study for subjects in prior VEGF Trap-Eye Phase I and II studies. Primary objective is to assess long-term safety and tolerability of continuing intravitreal treatment in subjects with wet age-related macular degeneration.

DETAILED DESCRIPTION:
Randomized, Single-Masked Phase II study for subjects previously enrolled in Phase I and II studies for wet age-related macular degeneration with VEGF Trap-Eye intravitreal injection as treatment.Long term (3 years) treatment is intended to measure safety and tolerability, as well as frequency of re-treatment and the effect of VEGF Trap-Eye on best corrected visual acuity (BCVA).

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in VEGF Trap-Eye Phase I and II studies

Exclusion Criteria:

* Any ocular or systemic adverse events that would preclude participation
* Presence of any condition that would jeopardize subject's participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2007-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (33):
- United States (33):
  - Peoria, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Loma Linda, California
  - Palm Springs, California
  - Pasadena, California
  - Poway, California
  - Westlake Village, California
  - Fort Myers, Florida
  - Stuart, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Glenview, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Boston, Massachusetts
  - West Springfield, Massachusetts
  - Toms River, New Jersey
  - Lynbrook, New York
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 35 sites in the United States that participated in the Phase 1 and Phase 2 studies VGFT OD-0502 (NCT00320775), -0508 (NCT00320788), or -0603 (NCT00383370). The recruitment period occurred between 19 Oct 2007 and 29 Oct 2008.
Pre-assignment Details: One hundred fifty seven participants were eligible if they had neovascular Age-related Macular Degeneration (AMD) and completed dosing in the Phase 1 and Phase 2 studies VGFT-OD-0502 (NCT00320775), -0508 (NCT00320788), or -0603 (NCT00383370). For each subject, only one eye was designated as the study eye.
Groups:
- Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg: The study consisted of a treatment period from day 1 to week 152, and a 4-week follow-up visit at week 156. Participants were scheduled to return to the clinical site every 8 weeks. At each visit, the investigator determined the need for an Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) based on his/her assessment of the participant (PRN or "as needed" dosing). If, at any point during the study, in the investigator's opinion, a participant required dosing or evaluation more frequently than every 8 weeks, monthly visits and dosing were permitted. The maximum frequency of injection into the study eye was every 4 weeks.
Period: Overall Study
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg
Started | 157
Completed | 120
Not Completed | 37
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 5
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 4
Not completed — OTHER | 4
Not completed — Death | 9

BASELINE CHARACTERISTICS:
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg
Number analyzed (Participants) | 157
Age Continuous [Mean (Standard Deviation); unit: years] | 77.9 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 153
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 156
  More than one race | 0
  Unknown or Not Reported | 0
Baseline Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: scores on a scale] — For BCVA, tested via the 4 meter ETDRS (Early Treatment Diabetic Retinopathy Study) protocol, 83 letter or more would represent 20/20 vision or better which would be considered an excellent outcome. Although, the ETDRS charts include 100 letters as the maximum possible score. The worst outcome is 0 letters read.
  scores on a scale | 61.3 (15.35)
Baseline Intraocular Pressure [Mean (Standard Deviation); unit: mmHg] — Intraocular pressure was measured in the study and fellow eyes using applanation tonometry or Tonopen at every study visit pre-dose, and 30 to 60 minutes post-injection.
  mmHg | 14.5 (3.12)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: Number of participants with AEs summarized by category
Time Frame: Baseline of this study to Wk 152
Measure: Number; unit: participants
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg
Number analyzed (Participants) | 157
participants
  Number of participants with any AE | 154
  Any ocular AE (Study eye and Fellow eye) | 138
  Any non ocular AE | 151
  Any treatment related AE (Ocular and non ocular) | 5
  Any SAE | 72
  Any AEs leading to withdrawal from study | 5
  Any Death due to AE | 11

2. Secondary Outcome: Frequency (Number of Injections)
Description: Frequency (number of injections) of PRN treatment from baseline of this study to week 152 (end of treatment).
Time Frame: Baseline of this study to Wk 152
Population: A total of 1116 PRN injections were administered into the study eyes of 135 participants between baseline of this study to Week 152 (end of treatment). Of the 157 enrolled participants, 22 received no injections, and 15 received 1 injection.
Measure: Median (Full Range); unit: Injections
Groups:
- Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg: The study consisted of a treatment period from day 1 to week 152 (end of treatment), and a 4-week follow-up visit at week 156 (end of study). Participants were scheduled to return to the clinical site every 8 weeks. At each visit, the investigator determined the need for an Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) based on his/her assessment of the participant (PRN or
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg
Number analyzed (Participants) | 157
Injections | 6.0 [0 to 26]

3. Secondary Outcome: Mean Change From Baseline of Original Study in Best Corrected Visual Acuity (BCVA) as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score of Study Eye - Observed Values
Description: Defined study baseline range of ETDRS Best Corrected Visual Acuity of: letter score of 73 to 25 (20/40 to 20/320) in the study eye; a higher score represents better functioning.
Time Frame: Baseline of original study to Wk 156
Measure: Mean (Standard Deviation); unit: letters read
Groups:
- Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg: The study consisted of a treatment period from day 1 to week 152, and a 4-week follow-up visit at week 156. Participants were scheduled to return to the clinical site every 8 weeks. At each visit, the investigator determined the need for an Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) based on his/her assessment of the participant (PRN or
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg
Number analyzed (Participants) | 157
letters read | 4.1 (17.71)

ADVERSE EVENTS:
Time Frame: Baseline of this study to Wk 156
Arm/Group | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg
Serious Adverse Events (participants affected / at risk) | 72/157
Other Adverse Events (participants affected / at risk) | 149/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg (N=157)
Anaemia (Blood and lymphatic system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Goitre (Endocrine disorders) | 1
Lens dislocation (Eye disorders) | 1 — Ocular AE Fellow Eye
Retinal oedema (Eye disorders) | 1 — Ocular AE Study Eye
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Gait disturbance (General disorders) | 1
Metaplasia (General disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 7
Atrioventricular block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Pericarditis (Cardiac disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Accident (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 — Ocular AE Study Eye
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Intraocular pressure increased (Investigations) | 1 — Ocular AE Fellow Eye
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Basal ganglia haemorrhage (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 2
Dementia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Hallucination (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Visual acuity reduced (Eye disorders) | 4 — Ocular AE Study Eye
Retinal haemorrhage (Eye disorders) | 2 — Ocular AE Study Eye
Cataract (Eye disorders) | 1 — Ocular AE Study Eye
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Aflibercept Injection (EYLEA, VEGF Trap-Eye) 2mg (N=157)
Anaemia (Blood and lymphatic system disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 12
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Hypertension (Vascular disorders) | 26
Age-related macular degeneration (Eye disorders) | 18 — Ocular AE Fellow Eye
Blepharitis (Eye disorders) | 13 — Ocular AE Fellow Eye
Cataract (Eye disorders) | 21 — Ocular AE Fellow Eye
Cataract nuclear (Eye disorders) | 9 — Ocular AE Fellow Eye
Conjunctival haemorrhage (Eye disorders) | 12 — Ocular AE Fellow Eye
Detachment of retinal pigment epithelium (Eye disorders) | 8 — Ocular AE Fellow Eye
Dry eye (Eye disorders) | 10 — Ocular AE Fellow Eye
Eye pain (Eye disorders) | 8 — Ocular AE Fellow Eye
Eye pruritus (Eye disorders) | 8 — Ocular AE Study Eye
Posterior capsule opacification (Eye disorders) | 10 — Ocular AE Study Eye
Retinal haemorrhage (Eye disorders) | 19 — Ocular AE Fellow Eye
Visual acuity reduced (Eye disorders) | 13 — Ocular AE Fellow Eye
Vitreous detachment (Eye disorders) | 11 — Ocular AE Fellow Eye
Vitreous floaters (Eye disorders) | 8 — Ocular AE Fellow Eye
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 16
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 14
Seasonal allergy (Immune system disorders) | 15
Bronchitis (Infections and infestations) | 17
Influenza (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 26
Sinusitis (Infections and infestations) | 16
Upper respiratory tract infection (Infections and infestations) | 24
Urinary tract infection (Infections and infestations) | 25
Contusion (Injury, poisoning and procedural complications) | 10
Fall (Injury, poisoning and procedural complications) | 29
Blood glucose increased (Investigations) | 13
Blood pressure increased (Investigations) | 9
Protein urine present (Investigations) | 13
White blood cell count increased (Investigations) | 12
White blood cells urine positive (Investigations) | 9
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 8
Depression (Psychiatric disorders) | 14
Insomnia (Psychiatric disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. There IS agreement between the Principal Investigator and the Sponsor that restricts the PI's rights to discuss or publish study results until Sponsor can review and comment. Sponsor can also remove confidential or proprietary information.